CLINICAL TRIAL: NCT05340569
Title: Diagnostic Value of Diffusion-weighted Magnetic Resonance Imaging for Detection of Peritoneal Metastases in High-risk Pancreatic Ductal Adenocarcinoma: a Pilot Study.
Brief Title: Diagnostic Value of DWI-MRI for Detection of Peritoneal Metastases in High-risk Pancreatic Ductal Adenocarcinoma.
Acronym: DWI-PDAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, Alexandre Brind'Amour, Doctor, Laval University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2022-6186
Record Dates: First submitted 2022-04-11; First posted 2022-04-22 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Pancreas Cancer, Duct Cell Adenocarcinoma; Pancreas Adenocarcinoma; Peritoneal Metastases; Peritoneal Carcinomatosis
Keywords: DWI; PDAC; Carcinomatosis; Diagnostic laparoscopy
MeSH Terms: conditions — Pancreatic Neoplasms; Peritoneal Neoplasms; Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- DWI-MRI (Experimental): Patients to undergo DWI-MRI (patients include in the study.
  Interventions: Diagnostic Test: Whole-body diffusion-weighted magnetic resonance imaging

INTERVENTIONS:
Diagnostic Test: Whole-body diffusion-weighted magnetic resonance imaging — See arm description.

SUMMARY:
Diffusion-weighted magnetic resonance imaging (DWI/MRI) has been described in recent literature as a highly sensitive and specific modality for the detection of peritoneal metastases (PM). It has been demonstrated to be superior to computed tomography (CT) for patients with known peritoneal disease from colorectal and gynaecological malignancies. However, the literature is scarce on the role of DWI/MRI in patients with pancreatic ductal-adenocarcinoma (PDAC). The aim of this study is to prospectively assess the added value of whole-body DWI/MRI (WB-DWI/MRI) to CT for detection of PM in the preoperative staging of patients with high-risk PDAC and evaluate how it correlates with intraoperative findings.

DETAILED DESCRIPTION:
This is a prospective study from a single center. Patients will be evaluated and operated on by one of five surgeons with a subspeciality in hepato-biliary and pancreatic surgery. After thorough assessment for resectability, patients with PDAC considered resectable based on CT, but at high-risk for peritoneal disease, will be prospectively included in the study and assessed with WB-DWI/MRI within 4 weeks of the planned surgery, with the standard protocol including the following sequences: Patients will drink 1L of pineapple juice one hour prior to the examination in order to provide a negative intraluminal contrast. Patients will receive 20 mg of intravenous hyoscine butylbromide at the beginning of the MR exam in order to reduce bowel peristalsis. Sequences will include Axial et Coronal T2WI of the abdomen and pelvis, axial DWI with b values of 0, 50 and 1000 of the abdomen and pelvis, as well as Pre and post gadolinium-based contrast Axial and Coronal 3D T1WGRE. Patients with no evidence of PM on WB-DWI/MRI will be operated on and undergo pancreatic resection following the usual exploration of the peritoneal cavity in case of occult metastatic disease. Patients with suspicion of PM on WB-DWI/MRI will be approached with a diagnostic laparoscopy first, then undergo pancreatic resection if no evidence of PM is found. Each case will be followed for at least 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of pancreatic ductal adenocarcinoma.
* Resectable disease or borderline resectable disease based on CT.
* Tumor size ≥ 3 cm.
* CA 19-9 ≥ 400 U/mL with normal bilirubin level (< 40)
* No evidence of distant metastases.
* Patient fit for pancreatic resection (ECOG 0 or 1).

Exclusion Criteria:

* Impossibility to obtain tissue diagnosis preoperatively confirming pancreatic ductal adenocarcinoma.
* Locally advanced disease on CT.
* Tumor size < 3 cm.
* CA 19-9 < 400 U/mL or CA 19-9 ≥ 400 U/mL with no preoperative drainage.
* Suspicion of distant metastases, including peritoneal metastases, on CT.
* Patient who is unable to have MRI.
* Patient unfit for pancreatic resection (ECOG 2 or more).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-03-28 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Peritoneal findings | 24 months
  The number of cases in which peritoneal findings on MRI altered clinical management.
Unexpected abortion | 24 months
  The rate of unexpected aborted surgery due to peritoneal metastases discovery at surgery.

SECONDARY OUTCOMES:
Early distant recurrence | 30 months
  The number of cases with early distant recurrence (less than 6 months).

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Brind'Amour, MD, Principal Investigator — Laval University
Locations (1):
- CHU de Québec, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Background] De La Cruz MS, Young AP, Ruffin MT. Diagnosis and management of pancreatic cancer. Am Fam Physician. 2014 Apr 15;89(8):626-32. PMID 24784121
- [Background] Hishinuma S, Ogata Y, Tomikawa M, Ozawa I, Hirabayashi K, Igarashi S. Patterns of recurrence after curative resection of pancreatic cancer, based on autopsy findings. J Gastrointest Surg. 2006 Apr;10(4):511-8. doi: 10.1016/j.gassur.2005.09.016. PMID 16627216
- [Background] Ryan DP, Hong TS, Bardeesy N. Pancreatic adenocarcinoma. N Engl J Med. 2014 Sep 11;371(11):1039-49. doi: 10.1056/NEJMra1404198. No abstract available. PMID 25207767
- [Background] Mizrahi JD, Surana R, Valle JW, Shroff RT. Pancreatic cancer. Lancet. 2020 Jun 27;395(10242):2008-2020. doi: 10.1016/S0140-6736(20)30974-0. PMID 32593337
- [Background] Patel CM, Sahdev A, Reznek RH. CT, MRI and PET imaging in peritoneal malignancy. Cancer Imaging. 2011 Aug 24;11(1):123-39. doi: 10.1102/1470-7330.2011.0016. PMID 21865109
- [Background] Allen VB, Gurusamy KS, Takwoingi Y, Kalia A, Davidson BR. Diagnostic accuracy of laparoscopy following computed tomography (CT) scanning for assessing the resectability with curative intent in pancreatic and periampullary cancer. Cochrane Database Syst Rev. 2016 Jul 6;7(7):CD009323. doi: 10.1002/14651858.CD009323.pub3. PMID 27383694
- [Background] Brind'Amour A, Webb M, Parapini M, Sideris L, Segedi M, Chung SW, Chartier-Plante S, Dube P, Scudamore CH, Kim PTW. The role of intraperitoneal chemotherapy in the surgical management of pancreatic ductal adenocarcinoma: a systematic review. Clin Exp Metastasis. 2021 Apr;38(2):187-196. doi: 10.1007/s10585-021-10074-2. Epub 2021 Jan 24. PMID 33486670
- [Background] Paracha M, Van Orden K, Patts G, Tseng J, McAneny D, Sachs T. Opportunity Lost? Diagnostic Laparoscopy in Patients with Pancreatic Cancer in the National Surgical Quality Improvement Program Database. World J Surg. 2019 Mar;43(3):937-943. doi: 10.1007/s00268-018-4855-8. PMID 30478680
- [Background] Jayakrishnan TT, Zacharias AJ, Sharma A, Pappas SG, Gamblin TC, Turaga KK. Role of laparoscopy in patients with peritoneal metastases considered for cytoreductive surgery and hyperthermic intraperitoneal chemotherapy (HIPEC). World J Surg Oncol. 2014 Aug 21;12:270. doi: 10.1186/1477-7819-12-270. PMID 25145962
- [Background] Vasilyeva E, Li J, Desai S, Chung SW, Scudamore CH, Segedi M, Kim PT. Impact of surgical wait times on oncologic outcomes in resectable pancreas adenocarcinoma. HPB (Oxford). 2020 Jun;22(6):892-899. doi: 10.1016/j.hpb.2019.10.013. Epub 2019 Nov 13. PMID 31732464
- [Background] Mattevi C, Garnier J, Marchese U, Ewald J, Gilabert M, Poizat F, Piana G, Delpero JR, Turrini O. Has the non-resection rate decreased during the last two decades among patients undergoing surgical exploration for pancreatic adenocarcinoma? BMC Surg. 2020 Aug 5;20(1):176. doi: 10.1186/s12893-020-00835-3. PMID 32758203
- [Background] Liu X, Fu Y, Chen Q, Wu J, Gao W, Jiang K, Miao Y, Wei J. Predictors of distant metastasis on exploration in patients with potentially resectable pancreatic cancer. BMC Gastroenterol. 2018 Nov 6;18(1):168. doi: 10.1186/s12876-018-0891-y. PMID 30400836
- [Background] De Rosa A, Cameron IC, Gomez D. Indications for staging laparoscopy in pancreatic cancer. HPB (Oxford). 2016 Jan;18(1):13-20. doi: 10.1016/j.hpb.2015.10.004. Epub 2015 Nov 18. PMID 26776846
- [Background] Dong L, Li K, Peng T. Diagnostic value of diffusion-weighted imaging/magnetic resonance imaging for peritoneal metastasis from malignant tumor: A systematic review and meta-analysis. Medicine (Baltimore). 2021 Feb 5;100(5):e24251. doi: 10.1097/MD.0000000000024251. PMID 33592867
- [Background] Dresen RC, De Vuysere S, De Keyzer F, Van Cutsem E, Prenen H, Vanslembrouck R, De Hertogh G, Wolthuis A, D'Hoore A, Vandecaveye V. Whole-body diffusion-weighted MRI for operability assessment in patients with colorectal cancer and peritoneal metastases. Cancer Imaging. 2019 Jan 7;19(1):1. doi: 10.1186/s40644-018-0187-z. PMID 30616608
- [Background] Zhang H, Dai W, Fu C, Yan X, Stemmer A, Tong T, Cai G. Diagnostic value of whole-body MRI with diffusion-weighted sequence for detection of peritoneal metastases in colorectal malignancy. Cancer Biol Med. 2018 May;15(2):165-170. doi: 10.20892/j.issn.2095-3941.2017.0162. PMID 29951340
- [Background] Namimoto T, Awai K, Nakaura T, Yanaga Y, Hirai T, Yamashita Y. Role of diffusion-weighted imaging in the diagnosis of gynecological diseases. Eur Radiol. 2009 Mar;19(3):745-60. doi: 10.1007/s00330-008-1185-5. Epub 2008 Oct 7. PMID 18839179
- [Background] De Vuysere S, Vandecaveye V, De Bruecker Y, Carton S, Vermeiren K, Tollens T, De Keyzer F, Dresen RC. Accuracy of whole-body diffusion-weighted MRI (WB-DWI/MRI) in diagnosis, staging and follow-up of gastric cancer, in comparison to CT: a pilot study. BMC Med Imaging. 2021 Feb 5;21(1):18. doi: 10.1186/s12880-021-00550-2. PMID 33546626